CLINICAL TRIAL: NCT02361515
Title: Moderate Hypofractionated Radiotherapy (62 Gy in 20 Fractions of 3.1 Gy) Versus Stereotactic Radiotherapy (37.5 Gy in 5 Fractions of 7.5 Gy) With Hyaluronic Acid Injection Between the Prostate and the Rectum for Prostate Cancer of Low- to Intermediate Risk; RPAH2
Brief Title: Hypofractionated Radiotherapy Versus Stereotactic Irradiation With Hyaluronic Acid
Acronym: RPAH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-846
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Adenocarcinoma
Keywords: Prostate; Hypofractionated radiotherapy; Stereotactic irradiation; Spacer; Rectal and bladder toxicities
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate Hypofractionated radiotherapy (62Gy) (Active Comparator): 20 fractions of 3.1Gy
  Interventions: Radiation: Moderate hypofractionated radiotherapy
- Stereotactic radiotherapy (37.5Gy) (Experimental): 5 fractions of 7.5Gy)
  Interventions: Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Radiation: Moderate hypofractionated radiotherapy — Moderate hypofractionated radiotherapy of 62Gy in 20 fraction of 3.1Gy.
  Arms: Moderate Hypofractionated radiotherapy (62Gy)
Radiation: Stereotactic radiotherapy — Stereotactic radiotherapy of 37.5Gy in 5 fraction of 7.5Gy.
  Arms: Stereotactic radiotherapy (37.5Gy)

SUMMARY:
The present randomized, open, multicentric Phase II trial, in parallel groups with two arms of treatment, compares the treatment A, moderate hypofractionated radiotherapy of 62Gy, to treatment B, stereotactic irradiation of 37.5 Gy with hyaluronic acid injection in the space between the prostate and the rectum to preserve the rectal-wall from high doses of irradiation. The study aims to assess the rates of late urinary toxicities of grade ≥ 2 induced by a moderate hypofractionated radiotherapy (62Gy in 20 fractions of 3.1Gy) and by a stereotactic radiotherapy (37.5Gy in 5 fractions of 7.5Gy), and the rectal toxicities after an injection of hyaluronic acid between the rectal wall and the prostate.

Ninety-six patients and 9 centers are included in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* age superior or equal to 18 years and inferior to 80 years.
* patient with a low- to intermediate-risk prostate cancer, according to D'Amico classification, for an exclusive irradiation.
* prostate cancer histologically proven.
* performance index OMS (World Health Organization) of grade 0-2.
* indication of external beam radiotherapy validate by the medical commission of the institution.
* IPSS (International Prostate Symptom Score < 15/35 (without alpha-blocker).
* the signed consent form.

Exclusion Criteria:

* Rectal surgery antecedents.
* prostate resection less than 6 mois.
* Involvement of the seminal vesicles or of the capsule on MRI.
* patient who can't cooperate during the treatment.
* pelvic irradiation antecedents.
* antecedents of inflammatory intestinal pathologies.
* neoplasia.
* patients treated with anti-neoplastic or anti-angiogenic or with other treatments used in rheumatology and which may include methotrexate (in order not to have a radiosensitizing effect).
* patients receiving anticoagulant treatment.
* other undergoing study that may interfere with the present study.
* patient under legal protection measure.
* hypersensitivity to hyaluronic acid.
* patient with auto-immune disease.
* patient receiving immunosuppressive medication.
* severe allergies.
* history of endocarditis.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with late urinary toxicities of grade ≥ 2 after moderate hypofractionated radiotherapy (62Gy in 20 fractions of 3.1Gy) and after stereotactic radiotherapy (37.5Gy in 5 fractions of 7.5Gy). | Follow-up at ≥ 3 months after the radiotherapy and up to 3 years.
  Late urinary toxicities of grade ≥ 2 assessed using the Common Toxicity Criteria for Adverse Effects ( CTCAE) v 4.0 classification from 3 months to 3 years.

SECONDARY OUTCOMES:
Survival rates without biological relapse in both arms. | 3 years.
  Survival rates without biological relapse (increase of the PSA (prostate-specific antigen) beyond nadir + 2 ng/ml, using Phoenix definition).
Evaluation and comparison of the acute urinary and rectal toxicities in both arms. | 3 months: evaluation at 3 months.
  all toxicities will be listed using Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0.
Evaluation and comparison of the sexual preservation rates in both arms. | 3 years.
  evaluation and comparison of the sexual preservation rates in both arms using International Index of Erectile Function (IIEF).
Late rectal toxicities in both arms, for the evaluation of the hyaluronic acid efficacy to preserve the rectal wall in both approaches. | 3 years.
  Late rectal toxicities in both arms, for the evaluation of the hyaluronic acid efficacy to preserve the rectal wall in both approaches, using Common Toxicity Criteria for Adverse Effects (CTCAE) 4.0.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Clinique Claude Bernard Service de radiothérapie CMCO Claude Bernard, Albi
  - Centre Georges Francois Leclerc, Dijon
  - Institut Paoli Calmettes, Marseille
  - Site Hospitalier Nord Boulevard Jacques Monod, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie de la Loire, Saint-Etienne
  - Groupe ONCORAD Clinique Pasteur, Toulouse

REFERENCES:
- [Derived] Jmour O, Benna M, Champagnol P, Ben Mrad M, Hamrouni A, Obeid L, Lahmamssi C, Bousarsar A, Vial N, Rehailia-Blanchard A, Sotton S, Lan M, Langrand-Escure J, Vallard A, Magne N. CBCT evaluation of inter- and intra-fraction motions during prostate stereotactic body radiotherapy: a technical note. Radiat Oncol. 2020 Apr 19;15(1):85. doi: 10.1186/s13014-020-01534-2. PMID 32307017